CLINICAL TRIAL: NCT00314951
Title: A Multi-National, Multi-Center, Double-Blind, Randomized, Parallel Group Study to Compare the Safety and Efficacy of 200 mg PAR-101 Taken q12h With 125 mg Vancomycin Taken q6h for Ten Days in Subjects With Clostridium Difficile-Associated Diarrhea
Brief Title: Fidaxomicin Versus Vancomycin for the Treatment of Clostridium Difficile-Associated Diarrhea (CDAD) (MK-5119-018)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Optimer Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5119-018; 101.1.C.003 (Other: Optimerpharma Study Number)
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Clostridium Infections; Diarrhea
Keywords: CDAD, Clostridium difficile, diarrhea; Clostridium difficile-Associated Diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — Fidaxomicin; OPT 80; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fidaxomicin (Experimental): Participants receiving fidaxomicin 200 mg capsules orally two times daily (every 12 hours [q12h] regimen) with intermittent matching placebo to fidaxomicin
  Interventions: Drug: Fidaxomicin; Drug: Matching Placebo to Fidaxomicin
- Vancomycin (Active Comparator): Participants receiving vancomycin 125 mg capsules orally four times daily (every 6 hours [q6h] regimen).
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Fidaxomicin — 200 mg oral capsules two times daily (q12h regimen)
  Other Names: PAR-101; OPT-80; Dificid®
  Arms: fidaxomicin
Drug: Vancomycin — 125 mg capsules q6hr (4 times a day)
  Arms: Vancomycin
Drug: Matching Placebo to Fidaxomicin — Matching Placebo to Fidaxomicin administered two times daily (intermittently with fidaxomicin dosing)
  Arms: fidaxomicin

SUMMARY:
This is a comparative study to investigate the safety and efficacy of fidaxomicin versus vancomycin in subjects with Clostridium difficile-Associated Diarrhea (CDAD).

DETAILED DESCRIPTION:
The primary objective of this pivotal study is to investigate the safety and efficacy of fidaxomicin versus vancomycin in subjects with Clostridium difficile-associated diarrhea (CDAD). The cure rates at end of therapy and recurrence rates will be evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Males/females with CDAD
* Females must use adequate contraception
* Signed informed consent

Exclusion Criteria:

* Life-threatening CDAD
* Toxic megacolon
* Pregnant
* Concurrent use of diarrheal agents
* Participation in other trials

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2006-05-02 (Actual); Primary Completion 2008-07-23 (Actual); Study Completion 2008-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Louie TJ, Miller MA, Mullane KM, Weiss K, Lentnek A, Golan Y, Gorbach S, Sears P, Shue YK; OPT-80-003 Clinical Study Group. Fidaxomicin versus vancomycin for Clostridium difficile infection. N Engl J Med. 2011 Feb 3;364(5):422-31. doi: 10.1056/NEJMoa0910812. PMID 21288078
- [Derived] D'Agostino RB Sr, Collins SH, Pencina KM, Kean Y, Gorbach S. Risk estimation for recurrent Clostridium difficile infection based on clinical factors. Clin Infect Dis. 2014 May;58(10):1386-93. doi: 10.1093/cid/ciu107. Epub 2014 Mar 5. PMID 24599770
- [Derived] Cornely OA, Miller MA, Fantin B, Mullane K, Kean Y, Gorbach S. Resolution of Clostridium difficile-associated diarrhea in patients with cancer treated with fidaxomicin or vancomycin. J Clin Oncol. 2013 Jul 1;31(19):2493-9. doi: 10.1200/JCO.2012.45.5899. Epub 2013 May 28. PMID 23715579
- [Derived] Cornely OA, Miller MA, Louie TJ, Crook DW, Gorbach SL. Treatment of first recurrence of Clostridium difficile infection: fidaxomicin versus vancomycin. Clin Infect Dis. 2012 Aug;55 Suppl 2(Suppl 2):S154-61. doi: 10.1093/cid/cis462. PMID 22752865
- [Derived] Louie TJ, Cannon K, Byrne B, Emery J, Ward L, Eyben M, Krulicki W. Fidaxomicin preserves the intestinal microbiome during and after treatment of Clostridium difficile infection (CDI) and reduces both toxin reexpression and recurrence of CDI. Clin Infect Dis. 2012 Aug;55 Suppl 2(Suppl 2):S132-42. doi: 10.1093/cid/cis338. PMID 22752862
- [Derived] Nerandzic MM, Mullane K, Miller MA, Babakhani F, Donskey CJ. Reduced acquisition and overgrowth of vancomycin-resistant enterococci and Candida species in patients treated with fidaxomicin versus vancomycin for Clostridium difficile infection. Clin Infect Dis. 2012 Aug;55 Suppl 2(Suppl 2):S121-6. doi: 10.1093/cid/cis440. PMID 22752860
- [Derived] Figueroa I, Johnson S, Sambol SP, Goldstein EJ, Citron DM, Gerding DN. Relapse versus reinfection: recurrent Clostridium difficile infection following treatment with fidaxomicin or vancomycin. Clin Infect Dis. 2012 Aug;55 Suppl 2(Suppl 2):S104-9. doi: 10.1093/cid/cis357. PMID 22752857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from May 2006 to August 2008 by centers in the United States and Canada.
Groups:
- Vancomycin: 125 mg administered 4 times daily (q6hr)
- Fidaxomicin: 200 mg administered twice daily (q12hr)
Period: Enrollment
Arm/Group | Vancomycin | Fidaxomicin
Started | 323 | 306
Completed | 323 (6 subjects took incorrect treatment assignment, 6 subjects didn't take drug) | 300 (6 subjects took incorrect treatment assignment, 6 subjects didn't take drug)
Not Completed | 0 | 6
Period: Treatment
Arm/Group | Vancomycin | Fidaxomicin
Started | 323 | 300
Completed | 307 | 289
Not Completed | 16 | 11
Not completed — Didn't meet criteria for mITT population | 16 | 11
Period: Follow-up
Arm/Group | Vancomycin | Fidaxomicin
Started | 307 | 289
Completed | 263 | 255
Not Completed | 44 | 34
Not completed — mITT failure | 44 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vancomycin | Fidaxomicin | Total
Number analyzed (Participants) | 307 | 289 | 596
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (16.9) | 60.3 (16.9) | 61.6 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 164 | 333
  Male | 138 | 125 | 263
Region of Enrollment [Number; unit: participants]
  United States | 186 | 165 | 351
  Canada | 121 | 124 | 245

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate at End of Therapy
Description: Percentage of participants with 3 or fewer unformed stools for 2 consecutive days and maintained through the end of therapy, and the subject no longer needed specific anti-Clostridium antibacterial treatment after completion of the course of study medication.
Time Frame: Study day 10 (+/- 2 days)
Population: Analysis data is modified intent to treat (mITT) population. The mITT population consists of subjects that had CDAD confirmed by >3 unformed bowel movements in the 24 hours prior to randomization and a positive toxin assay and received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vancomycin | Fidaxomicin
Number analyzed (Participants) | 307 | 289
Percentage of Participants | 85.7 [81.3 to 89.2] | 88.2 [84.0 to 91.5]
Statistical Analysis 1: Comparison: Vancomycin vs Fidaxomicin; H0: C(fidaxomicin) - C(Vancomycin) <= -10% Power calculation is based on cure rate of 85% in both treatment groups, non-inferiority margin of 10%, 2.5% (1-sided) type I error rate with approximately 90% power gives a total of 530 subjects; Test type: Non-Inferiority or Equivalence — The point estimate of the difference and the 2-sided 95% confidence interval (CI) for the difference between treatment groups were computed. If the lower limit of the CI was greater than -10%, the clinical non-inferiority of fidaxomicin was demonstrated. CIs for the difference of cure rates were calculated using the method recommended by Agresti and Caffo; Risk Difference (RD) = 2.6, 95% CI 2-sided [-2.9 to 8.0]

2. Secondary Outcome: Recurrence
Description: Percentage of participants with the re-establishment of diarrhea to an extent(based on frequency of passed unformed stools) that was greater than that noted on the last day of study medication, and the demonstration of either toxin A or B or both of C. difficile, and retreatment with CDI anti-infective therapy was needed.
Time Frame: Study days 11-40
Population: The mITT population for subjects who met the primary endpoint of cure subjects, were analyzed for the recurrence rates of diarrhea up to the Poststudy Visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vancomycin | Fidaxomicin
Number analyzed (Participants) | 263 | 255
Percentage of Participants | 25.1 | 15.7
Statistical Analysis 1: Comparison: Vancomycin vs Fidaxomicin; Test type: Superiority or Other; p = 0.008, Chi-squared; Risk Difference (RD) = -9.4, 95% CI 2-sided [-16.2 to -2.5]

3. Other Pre Specified Outcome: Global Cure
Description: Percentage of participants who were cured (3 or fewer unformed stools for 2 days through the end of therapy, and no C. difficile therapy after study drug completion) and didn't have recurrence (re-establishment of diarrhea that was greater than on the last day of study drug, positive C. difficile toxin and retreatment with C. difficile therapy) up to Day 40.
Time Frame: End of Study (Day 40)
Population: The analysis population is mITT, subjects that achieved a cure response at end of treatment and not having a recurrence at any time up to the Post-study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vancomycin | Fidaxomicin
Number analyzed (Participants) | 307 | 289
Percentage of Participants | 64.2 | 74.4
Statistical Analysis 1: Comparison: Vancomycin vs Fidaxomicin; Test type: Superiority or Other; p = 0.007, Chi-squared; Risk Difference (RD) = 10.2, 95% CI 2-sided [2.8 to 17.5]

ADVERSE EVENTS:
Time Frame: From Informed consent to 7-days following the last dose of study drug or until the last protocol-specified study visit, whichever occured later.
Arm/Group | Vancomycin | Fidaxomicin
Serious Adverse Events (participants affected / at risk) | 78/323 | 75/300
Other Adverse Events (participants affected / at risk) | 195/323 | 187/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vancomycin (N=323) | Fidaxomicin (N=300)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 4
Cardiogenic shock (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 3
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Cleft palate (Congenital, familial and genetic disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 4
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Megacolon (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Generalised oedema (General disorders) | 0 | 1
Hypothermia (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 6 | 3
Pneumonia (Infections and infestations) | 5 | 4
Sepsis (Infections and infestations) | 3 | 3
Staphylococcal bacteraemia (Infections and infestations) | 2 | 1
Staphylococcal sepsis (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 2 | 1
Aspergillosis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 2
Endocarditis bacterial (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pyelocystitis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Abdominal sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Fungaemia (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 1
Shunt infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Graft haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose abnormal (Investigations) | 1 | 1
Blood phosphorus decreased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 1 | 3
Lymphocyte count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood calcium increased (Investigations) | 0 | 1
Blood phosphorus abnormal (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Blood urea abnormal (Investigations) | 0 | 1
Blood uric acid abnormal (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal gland cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Mental status changes (Psychiatric disorders) | 3 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemopneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 2
Haemorrhage (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Vena cava thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vancomycin (N=323) | Fidaxomicin (N=300)
Anaemia (Blood and lymphatic system disorders) | 7 | 10
Nausea (Gastrointestinal disorders) | 28 | 31
Vomiting (Gastrointestinal disorders) | 14 | 18
Diarrhoea (Gastrointestinal disorders) | 12 | 9
Abdominal pain (Gastrointestinal disorders) | 7 | 9
Constipation (Gastrointestinal disorders) | 4 | 10
Oedema peripheral (General disorders) | 17 | 13
Pyrexia (General disorders) | 16 | 16
Chills (General disorders) | 8 | 1
Fatigue (General disorders) | 6 | 6
Pain (General disorders) | 5 | 6
Urinary tract infection (Infections and infestations) | 12 | 12
Pneumonia (Infections and infestations) | 8 | 6
Fall (Injury, poisoning and procedural complications) | 5 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 24 | 22
Dehydration (Metabolism and nutrition disorders) | 9 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 6
Headache (Nervous system disorders) | 14 | 20
Dizziness (Nervous system disorders) | 4 | 12
Insomnia (Psychiatric disorders) | 9 | 5
Renal failure acute (Renal and urinary disorders) | 2 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 9
Hypotension (Vascular disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less